CLINICAL TRIAL: NCT04947605
Title: Epidemiological Landscape of Cervical Cancer in Latin America .
Brief Title: Epidemiological Landscape of Cervical Cancer in Latin America
Acronym: EVITA LATAM
Status: Active, not recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 0820
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A portrait of clinical and epidemiological aspects of cervical cancer in Latin America is required to understand the high frequency of cervical cancer despite the existence of effective preventive tools. A better understanding of the current situation of this scenario will provide a valuable groundwork for the development of national and cooperative programs to improve cervical cancer prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years.
* Histologically proven cervical carcinoma
* Diagnosis of carcinoma of the cervix since January 2018 or newly diagnosis or recurrent disease during the period of study recruitment.
* Any histology of cervical cancer at time of diagnosis.
* FIGO stage IB2-IVA
* Have available and adequate medical records for data collection
* Accept to participate in the project and sign the informed consent (if applicable)

Exclusion Criteria:

* FIGO stage I and IB1
* Non-invasive cervical cancer
* Synchronous tumor or second primary tumor in the last five years (exception for thyroid cancer or skin cancer non melanoma)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from approximately 482 patients are planned to be collected in 7 (seven) countries in Latin America. Enrollment period for data collection is planned to be 18 months and follow-up data will be recorded for 5 years. Patients will receive treatment and clinical assessments for cervical cancer as determined by their treating physician, according to the standard of care and routine clinical practice at each site.
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
- Summarize the histologic subtype | January of 2028
  Summarize the histologic subtype, assessed by the anatomopathological assay of the tumor sample and the stage at diagnosis, assessed by FIGO stage (International Federation of Gynecology and Obstetrics (FIGO) staging of cancer of the cervix uteri - 2018), using gynecological exam. Image studies and TNM stage (AJCC 8th edition) will also be used to assess stage at diagnosis when available.

CONTACTS AND LOCATIONS:
Overall Officials: Graziela Zibetti Dal Molin, MD, Principal Investigator — Latin American Cooperative Oncology Group
Locations (1):
- A Real e Benemérita Associação Portuguesa de Beneficência, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Renna Junior NL, Silva GAE. Temporal trend and associated factors to advanced stage at diagnosis of cervical cancer: analysis of data from hospital based cancer registries in Brazil, 2000-2012. Epidemiol Serv Saude. 2018;27(2):e2017285. doi: 10.5123/s1679-49742018000200003. Epub 2018 May 7. English, Portuguese. PMID 29742234
- [Background] Nogueira-Rodrigues A. HPV Vaccination in Latin America: Global Challenges and Feasible Solutions. Am Soc Clin Oncol Educ Book. 2019 Jan;39:e45-e52. doi: 10.1200/EDBK_249695. Epub 2019 May 17. PMID 31099692
- [Background] Soneji S, Fukui N. Socioeconomic determinants of cervical cancer screening in Latin America. Rev Panam Salud Publica. 2013 Mar;33(3):174-82. doi: 10.1590/s1020-49892013000300003. PMID 23698136
- [Background] Lou H, Villagran G, Boland JF, Im KM, Polo S, Zhou W, Odey U, Juarez-Torres E, Medina-Martinez I, Roman-Basaure E, Mitchell J, Roberson D, Sawitzke J, Garland L, Rodriguez-Herrera M, Wells D, Troyer J, Pinto FC, Bass S, Zhang X, Castillo M, Gold B, Morales H, Yeager M, Berumen J, Alvirez E, Gharzouzi E, Dean M. Genome Analysis of Latin American Cervical Cancer: Frequent Activation of the PIK3CA Pathway. Clin Cancer Res. 2015 Dec 1;21(23):5360-70. doi: 10.1158/1078-0432.CCR-14-1837. Epub 2015 Jun 16. PMID 26080840
- [Background] Chung HC, Ros W, Delord JP, Perets R, Italiano A, Shapira-Frommer R, Manzuk L, Piha-Paul SA, Xu L, Zeigenfuss S, Pruitt SK, Leary A. Efficacy and Safety of Pembrolizumab in Previously Treated Advanced Cervical Cancer: Results From the Phase II KEYNOTE-158 Study. J Clin Oncol. 2019 Jun 10;37(17):1470-1478. doi: 10.1200/JCO.18.01265. Epub 2019 Apr 3. PMID 30943124
- [Background] Tewari KS, Sill MW, Long HJ 3rd, Penson RT, Huang H, Ramondetta LM, Landrum LM, Oaknin A, Reid TJ, Leitao MM, Michael HE, Monk BJ. Improved survival with bevacizumab in advanced cervical cancer. N Engl J Med. 2014 Feb 20;370(8):734-43. doi: 10.1056/NEJMoa1309748. PMID 24552320
- [Background] Cancer Genome Atlas Research Network; Albert Einstein College of Medicine; Analytical Biological Services; Barretos Cancer Hospital; Baylor College of Medicine; Beckman Research Institute of City of Hope; Buck Institute for Research on Aging; Canada's Michael Smith Genome Sciences Centre; Harvard Medical School; Helen F. Graham Cancer Center &Research Institute at Christiana Care Health Services; HudsonAlpha Institute for Biotechnology; ILSbio, LLC; Indiana University School of Medicine; Institute of Human Virology; Institute for Systems Biology; International Genomics Consortium; Leidos Biomedical; Massachusetts General Hospital; McDonnell Genome Institute at Washington University; Medical College of Wisconsin; Medical University of South Carolina; Memorial Sloan Kettering Cancer Center; Montefiore Medical Center; NantOmics; National Cancer Institute; National Hospital, Abuja, Nigeria; National Human Genome Research Institute; National Institute of Environmental Health Sciences; National Institute on Deafness &Other Communication Disorders; Ontario Tumour Bank, London Health Sciences Centre; Ontario Tumour Bank, Ontario Institute for Cancer Research; Ontario Tumour Bank, The Ottawa Hospital; Oregon Health &Science University; Samuel Oschin Comprehensive Cancer Institute, Cedars-Sinai Medical Center; SRA International; St Joseph's Candler Health System; Eli &Edythe L. Broad Institute of Massachusetts Institute of Technology &Harvard University; Research Institute at Nationwide Children's Hospital; Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University; University of Bergen; University of Texas MD Anderson Cancer Center; University of Abuja Teaching Hospital; University of Alabama at Birmingham; University of California, Irvine; University of California Santa Cruz; University of Kansas Medical Center; University of Lausanne; University of New Mexico Health Sciences Center; University of North Carolina at Chapel Hill; University of Oklahoma Health Sciences Center; University of Pittsburgh; University of Sao Paulo, Ribeir ao Preto Medical School; University of Southern California; University of Washington; University of Wisconsin School of Medicine &Public Health; Van Andel Research Institute; Washington University in St Louis. Integrated genomic and molecular characterization of cervical cancer. Nature. 2017 Mar 16;543(7645):378-384. doi: 10.1038/nature21386. Epub 2017 Jan 23. PMID 28112728